CLINICAL TRIAL: NCT01145625
Title: A Phase 3 Multi-Center Parallel Design Clinical Trial to Compare the Efficacy and Safety of 5 % Minoxidil Foam vs. 2 % Minoxidil Solution in Females for the Treatment of Female Pattern Hair Loss - Androgenetic Alopecia (MINALO3004, NCT01145625)
Brief Title: Clinical Trial in Females With Female Pattern Hair Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Healthcare Products Division of McNEIL-PPC, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MINALO3004; 2009-018109-29 (EudraCT Number)
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Alopecia
Keywords: Female Pattern Baldness
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5% MTF (Experimental): 5% Minoxidil Topical Foam
  Interventions: Drug: 5% Minoxidil
- 2% MTS (Active Comparator): 2% Minoxidil Topical Solution
  Interventions: Drug: 2% Minoxidil

INTERVENTIONS:
Drug: 5% Minoxidil — half a cap (equivalent to 1g) 5% Minoxidil Topical Foam applied to the scalp once daily, every day, for 52 weeks
  Arms: 5% MTF
Drug: 2% Minoxidil — one ml of 2% Minoxidil Topical Solution applied to the scalp two times a day, every day, for 52 weeks
  Other Names: ROGAINE®
  Arms: 2% MTS

SUMMARY:
This is a year-long clinical trial to evaluate the effectiveness and safety in women with Female Pattern Hair Loss (FPHL), comparing a new 5% minoxidil topical foam (MTF) formulation applied once a day versus the 2% minoxidil topical solution (MTS) applied twice a day.

This clinical trial uses an objective measurement called Target Area Hair Count (TAHC) to evaluate if there is a change in the number of hairs in the area being examined after using the product for 24 weeks (and also after using the product for 12 Weeks and for 52 weeks).

This trial will determine if the benefit of using either study product outweighs the risks.

DETAILED DESCRIPTION:
This is a phase 3, two-arm, randomized, active-controlled, multi-center, 52-week, parallel design trial to evaluate the efficacy and safety in women with Female Pattern Hair Loss (FPHL), comparing the new 5% minoxidil topical foam (MTF) formulation versus the 2% minoxidil topical solution (MTS) formulation.

This clinical trial is designed to compare the risk/benefit profile of the 5% MTF formulation applied once a day versus the 2% MTS applied twice a day (BID), using objective efficacy measures and safety assessments.

Study centers will screen a sufficient number of participants so that a minimum of 300 female participants with FPHL will be enrolled, to ensure 270 to complete. There will be at least 16 participants enrolled per center at multiple centers located across the US and globally. Approximately 300 participants will be randomly assigned in a 1:1 ratio to use either 5% MTF or 2% MTS, for 52 weeks for efficacy and safety evaluations.

Participants meeting the inclusion criteria will be randomly assigned in the order of their enrollment at each site. The signing of the informed consent and assignment of a participant number to a subject shall constitute enrollment.

During the trial following enrollment at Baseline, participants will return to the study site at regular intervals for safety assessments, adverse events monitoring, and compliance assessments. At the Week 12, 24, and Week 52 visits TAHC will be evaluated for efficacy analysis.

ELIGIBILITY:
Inclusion Criteria:

* females, age 18 or older in general good health
* exhibits female pattern hair loss
* signs and dates an informed consent document
* agrees to use an adequate method of birth control; if of childbearing potential
* shows a negative urine pregnancy test at Screening Visit
* is willing to maintain the same hair style, hair color, and hair regimen throughout the study
* is willing and able to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures

Exclusion Criteria:

* hypersensitivity to the study product, or any ingredients of the study product
* known allergy to hair dye, or hair dye components
* clinically relevant history of hypotension
* untreated or uncontrolled hypertension
* pregnant, planning a pregnancy or nursing a child
* history of hair transplants
* currently use hair weaves or non-breathable wigs
* dermatologic disorders of the scalp that require chronic use of medication for control
* other types or history of hair loss
* enrolled in any other investigational medication (drug) study currently, or within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Kendall, MA, Study Director — Johnson & Johnson Healthcare Products Division of McNEIL-PPC, Inc.
Locations (12):
- United States (8):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - University of Minnesota, Minneapolis, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Duke University Medical Center, Durham, North Carolina
  - NW Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, P.C., Portland, Oregon
  - DermResearch, Inc, Austin, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
- The Skin Care Centre, Vancouver, British Columbia, Canada
- Centre de Santé Sabouraud, Paris, Île-de-France Region, France
- Klinik für Dermatologie, Venerologie und Allergologie, Clinical Research Center for Hair and Skin Science, Berlin, Germany
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Blume-Peytavi U, Shapiro J, Messenger AG, Hordinsky MK, Zhang P, Quiza C, Doshi U, Olsen EA. Efficacy and Safety of Once-Daily Minoxidil Foam 5% Versus Twice-Daily Minoxidil Solution 2% in Female Pattern Hair Loss: A Phase III, Randomized, Investigator-Blinded Study. J Drugs Dermatol. 2016 Jul 1;15(7):883-9. PMID 27391640

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2% MTS | 5% MTF
Started | 161 | 161
Completed | 137 | 130
Not Completed | 24 | 31
Not completed — Lost to Follow-up | 8 | 9
Not completed — Adverse Event | 6 | 4
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 7 | 16
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population defined as all participants randomly assigned to a treatment group who received dispensed investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% MTS | 5% MTF | Total
Number analyzed (Participants) | 161 | 161 | 322
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 134 | 129 | 263
  >=65 years | 26 | 31 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 161 | 322
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 5 | 9
  White | 149 | 141 | 290
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Target Area Hair Count (TAHC)
Description: Number of hairs in the area being examined as measured by macrophotography.
Time Frame: Baseline to Week 24
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: hairs per centimeter squared
Arm/Group | 2% MTS | 5% MTF
Number analyzed (Participants) | 161 | 161
hairs per centimeter squared
  Baseline | 167.3 (55.0) | 169.7 (58.6)
  Week 24 | 192.8 (57.0) | 194.4 (64.7)
  Change from Baseline to Week 24 | 23.8 (24.7) | 23.7 (22.9)
Statistical Analysis 1: Comparison: 2% MTS vs 5% MTF; Statistical analysis is for the change from baseline to week 24 data; Test type: Non-Inferiority or Equivalence — Noninferiority was claimed if the lower limit of the 95% Confidence Interval (CI) was greater than -6.565; p = 0.9170, ANCOVA; P-Value and confidence interval are from ANCOVA model with treatment and center as factors and Baseline hair count as a covariate; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-6.0 to 5.4]

2. Secondary Outcome: Target Area Hair Count (TAHC)
Description: Number of hairs in the area being examined as measured by macrophotography
Time Frame: Baseline to Week 12
Population: Intent-to-Treat (ITT) population defined as all participants randomly assigned to a treatment group who received dispensed investigational product.
Measure: Mean (Standard Deviation); unit: hairs per centimeter squared
Arm/Group | 2% MTS | 5% MTF
Number analyzed (Participants) | 161 | 161
hairs per centimeter squared
  Baseline | 167.3 (55.0) | 169.7 (58.6)
  Week 12 | 190.7 (56.9) | 191.8 (62.6)
  Change from Baseline to Week 12 | 22.5 (22.8) | 24.9 (26.0)
Statistical Analysis 1: Comparison: 2% MTS vs 5% MTF; Statistical analysis is for the change from baseline to week 12 data; Test type: Superiority or Other; p < 0.4158, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-3.4 to 8.2]

3. Other Pre Specified Outcome: Target Area Hair Count (TAHC)
Description: Number of hairs in the area being examined as measured by macrophotography.
Time Frame: Baseline to Week 52
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: hairs per centimeter squared
Arm/Group | 2% MTS | 5% MTF
Number analyzed (Participants) | 161 | 161
hairs per centimeter squared
  Baseline | 167.3 (55.0) | 169.7 (58.6)
  Week 52 | 189.1 (55.8) | 186.9 (61.1)
  Change from Baseline to Week 52 | 19.4 (21.5) | 18.1 (23.4)
Statistical Analysis 1: Comparison: 2% MTS vs 5% MTF; Statistical analysis is for the change from baseline to week 52 data; Test type: Superiority or Other; p = 0.5980, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-7.1 to 4.1]

ADVERSE EVENTS:
Arm/Group | 2% MTS | 5% MTF
Serious Adverse Events (participants affected / at risk) | 8/161 | 2/161
Other Adverse Events (participants affected / at risk) | 118/161 | 109/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2% MTS (N=161) | 5% MTF (N=161)
Anal Abscess (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2% MTS (N=161) | 5% MTF (N=161)
Nasopharyngitis (Infections and infestations) | 22 | 23
Upper respiratory tract infection (Infections and infestations) | 8 | 16
Sinusitis (Infections and infestations) | 12 | 10
Urinary tract infection (Infections and infestations) | 3 | 8
Bronchitis (Infections and infestations) | 2 | 8
Cystitis (Infections and infestations) | 4 | 4
Gastroenteritis (Infections and infestations) | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Procedural pain (Injury, poisoning and procedural complications) | 6 | 4
Fall (Injury, poisoning and procedural complications) | 3 | 4
Weight increased (Investigations) | 14 | 20
Headache (Nervous system disorders) | 16 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Toothache (Gastrointestinal disorders) | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Influenza like illness (General disorders) | 3 | 4
Hypertension (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Multi-Center Publication will be the first publication to present the results of the Study. Upon such Multi-Center Publication, or the earlier of (a) Sponsor's confirmation that there will be no Multi-Center Publication or presentation, or (b) 12 months after the completion of the entire multi-center study, Institution and Investigator may publish or present Study data and results generated in their performance of the Study in accordance with the terms of this Article.